CLINICAL TRIAL: NCT03434054
Title: The Effect of Losartan on Emotional Processing in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MSD-IDREC-C3-2015-832
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
Keywords: losartan; emotional processing; anxiety; magnet resonance imaging; MRI
MeSH Terms: conditions — Anxiety Disorders | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled experimental medicine study, where healthy volunteers are randomised to receiving either a single dose of losartan (50mg) or matching placebo.
Who Masked: Participant, Investigator
Masking Description: Study medication and placebo are over-encapsulated to look identical, and both the participants and investigators in direct contact with partiicpants are blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan (Experimental): single dose of 50mg losartan, tablet, over-encapsulated, to be taken orally
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): single dose of placebo (main ingredient microcrystalline cellulose), tablet, over-encapsulated, to be taken orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan — blood pressure medication
  Other Names: Losartan Potassium
  Arms: Losartan
Other: Placebo — non-active sham intervention
  Arms: Placebo

SUMMARY:
This experimental medicine study explores whether a single dose of losartan (50mg) versus placebo affects the processing of positive and negative stimuli, using fMRI.

DETAILED DESCRIPTION:
Losartan has been shown to accelerate fear extinction in animals and to prevent the development of anxiety disorders in humans, emphasising its potential to possibly enhance exposure therapy in humans. This study explores the basic effects of losartan on emotional processing, to identify neural mechanisms by which the drug might have synergistic effects on psychological treatment in humans.

In a double-blind between-groups design, 30 healthy volunteers will be randomised to a group receiving a single dose of losartan (50mg) versus placebo, and this study will measure the effects of probing renin-angiotensin function on emotional information processing, using functional magnet resonance imaging (fMRI). Such knowledge will ultimately be essential for the development of more effective pharmaco-psychological treatment approaches for anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide informed consent
* male or Female, aged 18-50
* body mass index (BMI) of 18-30 kg/m2
* fluent English skills
* non- or light-smoker (< 5 cigarettes a day)

Exclusion Criteria:

* Female participant who is pregnant or breast-feeding
* central nervous system (CNS) active medication during the last 6 weeks
* Current blood pressure/other heart medication (esp. aliskiren or beta blockers)
* Intravascular fluid depletion
* Past or present DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) axis-I diagnosis
* Alcohol or substance abuse
* First-degree family member with a history of a severe psychiatric disease
* Impaired liver or kidney function
* Lifetime history of epilepsy or other neurological disease, systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Insufficient English skills
* participated in another study involving certain medication during last 6 weeks
* Contraindication to magnet resonance imaging (MRI) scanning (e.g. pacemaker)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
BOLD signal change | 1 day
  BOLD signal change during functional magnet resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Study Chair — University of Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reinecke A, Browning M, Klein Breteler J, Kappelmann N, Ressler KJ, Harmer CJ, Craske MG. Angiotensin Regulation of Amygdala Response to Threat in High-Trait-Anxiety Individuals. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Oct;3(10):826-835. doi: 10.1016/j.bpsc.2018.05.007. Epub 2018 Jun 5. PMID 29980493